CLINICAL TRIAL: NCT01440387
Title: A Phase IIIA Study of Immunogenicity and Safety of GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine FLU-Q-QIV in Adults Aged 18 Years and Older
Brief Title: A Study of Immunogenicity and Safety of GSK Biologicals' Influenza Vaccine FLU-Q-QIV in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115418
Record Dates: First submitted 2011-09-08; First posted 2011-09-26 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Influenza; Phase III; Seasonal influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- FLULAVAL QUADRIVALENT Adult Group (Experimental): Subjects 18-60 years of age received 1 dose of FLULAVAL® QUADRIVALENT vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: FLULAVAL® QUADRIVALENT
- FLULAVAL QUADRIVALENT Elderly Group (Experimental): Subjects above 60 years of age received 1 dose of FLULAVAL® QUADRIVALENT vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: FLULAVAL® QUADRIVALENT

INTERVENTIONS:
Biological: FLULAVAL® QUADRIVALENT — Intramuscular injection, 1 dose each in FLULAVAL QUADRIVALENT Adults and FLULAVAL QUADRIVALENT Elderly Groups

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of GlaxoSmithKline (GSK) Biologicals' investigational quadrivalent split virion influenza vaccine FLU-Q-QIV in adults 18 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject
* Male and female adults, 18 years of age and older in stable health as determined by investigator's clinical examination and assessment of subjects' medical history.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination

Exclusion Criteria:

* Administration of any influenza vaccine within 6 months preceding the study start or planned use of such vaccines during the study period.
* Administration of any other vaccine(s) within 30 days prior to study enrolment or during the study period.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Acute disease and/or fever at the time of enrolment.
* Significant acute or chronic, uncontrolled medical or psychiatric illness.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, based on history and physical examination.
* Insulin-dependent diabetes mellitus.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to study vaccine dose.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* History of chronic alcohol abuse and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g. low-dose aspirin, and without a clinically apparent bleeding tendency are eligible
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of FLU-Q-QIV and/or a history of anaphylactic type reaction to consumption of eggs, and/or reactions to products containing mercury.
* A history of severe adverse reaction to a previous influenza vaccination.
* Pregnant and/or lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-09-30; Primary Completion 2011-10-22 (Actual); Study Completion 2011-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jain VK, Chandrasekaran V, Wang L, Li P, Liu A, Innis BL. A historically-controlled Phase III study in adults to characterize the acceptability of a process change for manufacturing inactivated quadrivalent influenza vaccine. BMC Infect Dis. 2014 Mar 10;14:133. doi: 10.1186/1471-2334-14-133. PMID 24606983
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115418 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Started | 56 | 56
Completed | 56 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (13.33) | 68.6 (4.72) | 54.75 (17.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Hemagglutination Inhibition (HI) Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: Antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu B/Florida/4/06 (Yamagata), FluB/Bri/60/08 (Victoria), Flu A/CAL/7/09 (H1N1) and Flu A/Victoria/210/09 (H3N2) antigens.
Time Frame: At Day 0 and Day 21
Population: The analyses were performed on According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. These included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Titers
  Yamagata strain, Day 0 | 130.4 [92.8 to 183.2] | 57.3 [44.3 to 74.0]
  Yamagata strain, Day 21 | 404.8 [323.1 to 507.2] | 355.5 [263.5 to 479.5]
  Victoria strain, Day 0 | 92.8 [66.5 to 129.4] | 38.5 [28.3 to 52.4]
  Victoria strain, Day 21 | 318.0 [251.4 to 402.3] | 237.8 [179.7 to 314.9]
  H1N1 strain, Day 0 | 82.0 [54.9 to 122.5] | 25.0 [17.3 to 36.0]
  H1N1 strain, Day 21 | 392.5 [305.4 to 504.4] | 223.5 [157.0 to 318.1]
  H3N2 strain, Day 0 | 45.3 [31.3 to 65.4] | 23.2 [16.4 to 32.8]
  H3N2 strain, Day 21 | 215.4 [166.3 to 278.9] | 160.1 [115.7 to 221.4]

2. Primary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection. The vaccine strains assessed were Yamagata, Victoria, H1N1 and H3N2 antigens.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  Yamagata strain, Day 0 | 48 | 45
  Yamagata strain, Day 21 | 56 | 56
  Victoria strain, Day 0 | 47 | 31
  Victoria strain, Day 21 | 56 | 55
  H1N1 strain, Day 0 | 44 | 26
  H1N1 strain, Day 21 | 55 | 52
  H3N2 strain, Day 0 | 34 | 28
  H3N2 strain, Day 21 | 54 | 53

3. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Yamagata, Victoria, H1N1 and H3N2 antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  Yamagata strain | 20 | 35
  Victoria strain | 19 | 33
  H1N1 strain | 28 | 34
  H3N2 strain | 27 | 35

4. Primary Outcome: HI Antibody Seroconversion Factors (SCFs) Against Each of the 4 Vaccine Influenza Strains.
Description: SCFs were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains assessed were Yamagata, Victoria, H1N1 and H3N2 antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Fold increase
  Yamagata strain | 3.1 [2.4 to 4.0] | 6.2 [4.6 to 8.4]
  Victoria strain | 3.4 [2.5 to 4.6] | 6.2 [4.3 to 8.8]
  H1N1 strain | 4.8 [3.3 to 7.0] | 8.9 [5.8 to 13.7]
  H3N2 strain | 4.8 [3.5 to 6.6] | 6.9 [4.7 to 10.1]

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 redness and swelling were defined as redness/swelling greater than 100 millimeters (mm). i.e. >100mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  Any Pain | 41 | 19
  Grade 3 Pain | 0 | 0
  Any Redness | 1 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 1 | 2
  Grade 3 Swelling | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were chest tightness, chills, cough, fatigue, headache, joint pain at other location, muscle pain, red eyes, sore throat, swelling of the face and fever [oral temperature ≥ 38.0 degrees Celsius (°C)]. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = oral temperature above 39.0°C
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  Any Chest tightness | 0 | 2
  Grade 3 Chest tightness | 0 | 0
  Related Chest tightness | 0 | 2
  Any Chills | 1 | 5
  Grade 3 Chills | 0 | 0
  Related Chills | 1 | 5
  Any Cough | 3 | 4
  Grade 3 Cough | 0 | 0
  Related Cough | 3 | 4
  Any Fatigue | 10 | 5
  Grade 3 Fatigue | 0 | 1
  Related Fatigue | 10 | 5
  Any Headache | 11 | 5
  Grade 3 Headache | 0 | 0
  Related Headache | 11 | 5
  Any Joint pain at other location | 7 | 3
  Grade 3 Joint pain at other location | 0 | 0
  Related Joint pain at other location | 7 | 3
  Any Muscle pain | 21 | 6
  Grade 3 Muscle pain | 0 | 1
  Related Muscle pain | 21 | 6
  Any Red eyes | 3 | 0
  Grade 3 Red eyes | 0 | 0
  Related Red eyes | 3 | 0
  Any Sore throat | 7 | 5
  Grade 3 Sore throat | 0 | 0
  Related Sore throat | 7 | 5
  Any Swelling of the face | 0 | 0
  Grade 3 Swelling of the face | 0 | 0
  Related Swelling of the face | 0 | 0
  Any Fever | 0 | 0
  Grade 3 Fever | 0 | 0
  Related Fever | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period.
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects | 13 | 12

8. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Day 20 after vaccination).
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: During the entire study period (Days 0 - 20 after vaccination); Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 21-day (Days 0-20) post-vaccination period.
Description: For the systematically and non-systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | FLULAVAL QUADRIVALENT Adult Group | FLULAVAL QUADRIVALENT Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 46/56 | 28/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FLULAVAL QUADRIVALENT Adult Group (N=56) | FLULAVAL QUADRIVALENT Elderly Group (N=56)
Pain (General disorders) | 41 | 19
Chills (General disorders) | 1 | 5
Cough (General disorders) | 3 | 4
Fatigue (General disorders) | 10 | 5
Headache (General disorders) | 11 | 5
Joint pain at other location (General disorders) | 7 | 3
Muscle pain (General disorders) | 21 | 6
Red eyes (General disorders) | 3 | 0
Sore throat (General disorders) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.